CLINICAL TRIAL: NCT04943770
Title: Prospective Single-centre, Double-blind, Randomised Study to Evaluate the Effect of Spinal Cord Stimulation Frequency on wash-in/Wash-out Time and Clinical Outcomes in Subjects Using Fast-Acting Sub-perception Therapy (FAST) for Chronic Pain
Brief Title: Evaluating the Effect of Spinal Cord Stimulation Frequency on Fast-Acting Sub-perception Therapy (FAST) for Chronic Pain
Acronym: CHRONOS
Status: Withdrawn | Type: Observational
Why Stopped: COVID
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 281237
Record Dates: First submitted 2020-04-03; First posted 2021-06-29 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Neuropathic Low Back Pain
Keywords: spinal cord stimulation; sub-perception; low back pain; wash in/wash out; neuropathic pain
MeSH Terms: conditions — Low Back Pain; Neuralgia | interventions — Spinal Cord Stimulation; Drug Delivery Systems

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- WaveWriter™ Alpha Spinal Cord Stimulator (SCS) system: Patients will be randomised 4:4 to a specific stimulating rates order (A, B, C, D) for approx. 3-6 weeks per rate (12-24 weeks in total). Each period is followed by a wash-out phase.
  At each frequency systematic assessment of the sweet-spot(s) will be performed. Various pulse width and amplitude values may be used to optimize therapy (up to 1KHz). These programmes will be saved in the subject's remote control based on the pre-generated rate randomization sequence.
  Interventions: Procedure: Spinal cord stimulator implant; Diagnostic Test: Healing period; Device: WaveWriter™ Alpha Spinal Cord Stimulator (SCS) system

INTERVENTIONS:
Procedure: Spinal cord stimulator implant — Patients will undergo spinal cord implant procedures as per standard of care and be implanted with the WaveWriter™ Alpha Spinal Cord Stimulator (SCS) system.
  Implant Procedures will be followed by a healing period (4-6 weeks) during which patients will be offered therapy (up to one 1Khz). Patients will then be randomised to receive therapy at four different rates (A, B, C, D) in no particular order for 3-6 weeks each. Patients will then be followed up at 3 and 6 months after the last randomization visit.
  Other Names: Boston Scientific Wavewriter
Diagnostic Test: Healing period — Acute opioid pain medications may be continued. No additional scheduled assessments will be completed during this period.
Device: WaveWriter™ Alpha Spinal Cord Stimulator (SCS) system — Patients will then be randomised to receive therapy (up to 1KHz) at four different rates in no particular order for 3-6 weeks each. Patients will then be followed up at 3 and 6 months after the last randomization visit.

SUMMARY:
The study design is prospective, post-market, exploratory, single-centre, rate randomised, double-blinded (subject, evaluator blinded; programmer un-blinded). The study is designed to evaluate the wash-in and wash-out time of FAST (Fast Acting Sub-perception Therapy) at 90 Hz and various frequencies above and below 90 Hz.

A prospective study design will eliminate the bias associated with case selection in a retrospective review and will ensure that identical procedures are followed for data capture and review.

Randomization of rates will be used to minimise the sequence effects and the impact of carryover effects, as well as addressing issues that may be related to order effect.

The electronic diary will be used to log the subjects' pain intensity and medication usage. Additionally, the numerical rating scale for measuring pain intensity is a validated measure and has been used in other randomized controlled trials to measure the outcomes of spinal cord stimulation (SCS).

The electronic real-time NRS (Numerical rating score) recording will be used to log the subjects' pain intensity and time during wash-in evaluation session.

This study aims to evaluate pain relief and wash-in/wash-out frequency sensitivity using FAST at different stimulation rates. The different randomization period included in the study design allows for comparing these treatments using one of the stimulation rates as an active control.

DETAILED DESCRIPTION:
Chronic Pain Background

Chronic intractable pain is a significant worldwide health issue, which consumes considerable healthcare resources and heavily impacts the quality of life for many patients. It is often defined as pain persisting for at least 6 months and not responding to conservative treatment(s). Chronic pain may be induced by current or past nerve injury and causes significant disability. People affected by such condition often experience reduced health-related quality of life, reduced ability to engage in activities of daily living, depression, sleep disturbances and weight gain due to the adoption of a sedentary lifestyle.

Typical entry into the pain management continuum includes over-the-counter medications, followed by physical therapy and complementary medicine. Interventional Pain management, Interdisciplinary pain management and surgery are attempted next and are often followed by long-term oral opioids intake. Active implantable options, including Spinal Cord Stimulation (SCS), lie within the continuum of chronic pain therapies and can be recommended as an alternative to long-term opioids intake (as recommended by National Institute of Clinical Excellence- NICE).

Spinal Cord Stimulation (SCS)

SCS refers to the application of small amounts of electrical energy, often via wires (a.k.a. "leads") to stimulate nerves in the spinal cord and reduce chronic pain symptoms. SCS is a less invasive treatment option for chronic pain that has generally been reserved for patients who have failed multiple, and sometimes all, conservative chronic pain therapies. With SCS, an implanted pulse generator (IPG) delivers electrical current to leads implanted in the epidural space at specific spinal level. Electrical currents stimulates nerves and can be shaped to optimise stimulation of fibres innervating the painful locations, thereby reducing pain sensation.

For decades, paresthesia-based SCS has been used to treat chronic pain. The classic approach typically uses frequencies between 40-100 Hz and enables a relatively straightforward identification and energy-efficient stimulation of the so-called therapeutic "sweet-spot". However, a potential drawback of this method of treatment is that patients using paresthesia-based SCS must endure paresthesias ("tingling") which, although may not always be bothersome and even pleasant to some, is an aspect that some may prefer to avoid.

Although, within the last 10 years, SCS device technologies have expanded considerably. One example is the introduction of higher stimulation frequency (i.e., 10 kHz) and amplitudes below perception threshold, enabling patients to obtain pain relief without experiencing paresthesia. This approach is known as sub-perception SC. However, this method is very energy-intensive, requires patients to recharge every 1-2 days and exhibits a slow "wash-in" time (i.e., the time between therapy activation and relief from pain). Conventional sub-perception methodologies have the desirable property of not requiring the patient to feel paresthesia but have some notable drawbacks. In particular, (1) patients leave the clinic still awaiting relief and hoping that one of the programs provided will be effective, (2) the sweet-spot is assessed via a "blind" search, an approach that limits the number of program settings testable on each patient and calling into question whether or not the final settings are optimal, (3) and in many cases the programs require much more energy than a paresthesia-based program.

As part of an effort to improve patients' experience and outcomes associated with the utilization of sub-perception SCS, the investigators hypothesised that there might be a putative relationship between the following: a) the specific location in which a sub-perception stimulation field is most effective and b) the paresthesia that overlaps the physical area(s) of pain as reported by each patient. Evaluation of this hypothesis led the investigators to develop a novel approach for implementation of sub-perception SCS, which is termed "Fast Acting Sub-perception Therapy" (FAST). This new methodology offers all the advantages provided by both paresthesia- and sub-perception-based SCS while simultaneously mitigating the potential downsides typically associated with each of these modalities when they are applied independently.

Study objectives and Endpoints

Primary objective

The primary objective of this study is to evaluate the wash-in/wash-out times of Fast-Acting Sub-perception Therapy (FAST) and best clinical outcomes as measured by mean reported pain on Numerical Rating Scale at 90 Hz and with frequencies above and below 90 Hz.

Secondary objective

The secondary objective will be to investigate the effect on functionality, quality of life, therapy longevity (3 and 6-month) and adverse events in the study population.

Primary endpoint

There are no Primary Endpoints for this exploratory study.

Exploratory endpoint

The following exploratory endpoints will be collected in this study:

* Wash-in time of overall pain intensity (RT-NRS) of each Rate Randomization (A, B, C, D)
* Wash-out time of lower back, legs pain and overall pain intensity (ED-NRS) of each Rate Randomization (A, B, C, D)
* Change in average lower back, legs pain and overall pain intensity (ED-NRS) from Baseline to end of each Randomization (A, B, C, D) and Long-Term Follow-up periods
* Treatment Satisfaction at end of each Rate Randomization (A, B, C, D) and Long-Term Follow-up periods (PSWT)
* Global impression of change at end of each Rate Randomization (A, B, C, D) and Long-Term Follow-up periods (PGIC)
* Change in disability from Baseline to end of each Rate Randomization (A, B, C, D) and Long-Term Follow-up periods (ODIv2.1a)
* Change in Quality of life from Baseline to end of each Rate Randomization (A, B, C, D) and Long-Term Follow-up periods (EQ-5D-5L)
* Change in sleep quality from Baseline to end of each Rate Randomization (A, B, C, D) and Long-Term Follow-up periods (PSQ3)
* Subject preferred program at Long-Term Follow-up period (Preference Questionnaire)
* Pain/paresthesia overlap for each tested configuration at Rate Randomization (A, B, C, D) and Long-Term Follow-up periods (Pain/Paresthesia drawing

ELIGIBILITY:
Inclusion Criteria:

* The subject is between 18 and 75 years of age when written informed consent is obtained.
* Complaint of persistent or recurrent low back pain, with or without equal or lesser leg pain, for at least 90 days prior to Screen.
* Received at least 90 days of documented pain management care to address the primary pain complaint, prior to Screening (e.g. medication, physical therapy.)
* Diagnosed with chronic neuropathic pain of the low back and legs (of neuropathic origin only).
* Eligible candidate for SCS from a psychological and psychiatric standpoint as determined prior to Baseline Visit, per site's routine screening process No back surgery within 6 months prior to Screening.
* Average low back pain intensity, during the position/activity, which routinely causes worst pain, of 5 or greater on a 0-10 numerical rating scale during Baseline period based on eDiary.
* If taking prescription opioids for primary chronic pain complaint (low back and/or leg pain), must have been on a stable prescription (same drug(s) and dose(s)) 30 days prior to Screening to a total of less than 180 mg Oral Morphine equivalent.
* Willing and able to comply with all protocol-required procedures and assessments/evaluations (e.g. willing to comply with opioid prescription lock from the Baseline visit through End of Rate Randomization and protocol required stimulation parameter locks, complete daily eDiary).
* If female of childbearing potential: not pregnant, as evidenced by a negative pregnancy test at Screening.
* Subject signed a valid, IRB-approved informed consent form (ICF) provided in English.

Exclusion Criteria:

* Significant cognitive impairment at Screening that, in the opinion of the Investigator, would reasonably be expected to impair the study candidates to participate in the study
* Have untreated major psychiatric comorbidity, serious drug related behaviour issues.
* Previous spinal cord stimulation trial or is already implanted with an active implantable device(s) (e.g. pacemaker, drug pump, implantable pulse generator).
* Participating (or intends to participate) in another drug or device clinical trial that may influence the data that will be collected for this study
* Currently on any anticoagulant medications that cannot be discontinued during perioperative period
* Current condition associated with risk of immunocompromised that might increase risk of infection during study duration.
* A female who is pregnant, is breastfeeding, or is of childbearing potential and planning to get pregnant during the study or not using adequate contraception.
* Primary pain complaint of vascular origin (e.g. peripheral vascular disease). Spinal pain secondary to neoplasm, infection, autoimmune disorder with spinal involvement, or a spinal metabolic disorder.
* Clinically significant lumbosacral stenosis which would interfere with lead placement
* Prior history of lumbar-sacral spine fusion
* Any pain-related diagnosis or medical/psychological condition that, in the clinician's best judgment might confound reporting of study outcomes (e.g. pelvic pain, angina pain, chronic migraine.
* Radiographic evidence of spinal instability requiring fusion
* Terminal illness with anticipated survival 1 year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from neuropathic back pain with or without additional neuropathic leg pain that have not received any benefit from conventional medical management.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating scale | Baseline- patient visit at start of the study
  NRS will be used to measure the pain intensity, enabling the patient to express the severity of pain by giving it a numerical value from 0 to 10 on an 11-point numerical pain rating scale with 0 being no pain at all and 10 being the worst pain imaginable. An average overall score, back pain score, and leg pain score will be recorded.
Numerical Rating scale for Randomisation Arm A | up to 6 weeks
  NRS will be used to measure the pain intensity, enabling the patient to express the severity of pain by giving it a numerical value from 0 to 10 on an 11-point numerical pain rating scale with 0 being no pain at all and 10 being the worst pain imaginable. An average overall score, back pain score, and leg pain score will be recorded.
Numerical Rating scale for Randomisation Arm B | up to 6 weeks
  NRS will be used to measure the pain intensity, enabling the patient to express the severity of pain by giving it a numerical value from 0 to 10 on an 11-point numerical pain rating scale with 0 being no pain at all and 10 being the worst pain imaginable. An average overall score, back pain score, and leg pain score will be recorded.
Numerical Rating scale for Randomisation Arm C | up to 6 weeks
  NRS will be used to measure the pain intensity, enabling the patient to express the severity of pain by giving it a numerical value from 0 to 10 on an 11-point numerical pain rating scale with 0 being no pain at all and 10 being the worst pain imaginable. An average overall score, back pain score, and leg pain score will be recorded.
Numerical Rating scale for Randomisation Arm D | up to 6 weeks
  NRS will be used to measure the pain intensity, enabling the patient to express the severity of pain by giving it a numerical value from 0 to 10 on an 11-point numerical pain rating scale with 0 being no pain at all and 10 being the worst pain imaginable. An average overall score, back pain score, and leg pain score will be recorded.
Numerical Rating scale | 3 months post-randomisation
  NRS will be used to measure the pain intensity, enabling the patient to express the severity of pain by giving it a numerical value from 0 to 10 on an 11-point numerical pain rating scale with 0 being no pain at all and 10 being the worst pain imaginable. An average overall score, back pain score, and leg pain score will be recorded.
Numerical Rating scale | 6 months post randomisation
  NRS will be used to measure the pain intensity, enabling the patient to express the severity of pain by giving it a numerical value from 0 to 10 on an 11-point numerical pain rating scale with 0 being no pain at all and 10 being the worst pain imaginable. An average overall score, back pain score, and leg pain score will be recorded.
Oswestry Disability Index (ODI) | Baseline
  Oswestry Disability Index is a commonly used scale for back pain subjects with a neuropathic pain component. The test is considered the 'gold standard' of low back functional outcome tools.
Oswestry Disability Index (ODI) for Randomisation Arm A | up to 6 weeks
  Oswestry Disability Index is a commonly used scale for back pain subjects with a neuropathic pain component. The test is considered the 'gold standard' of low back functional outcome tools.
Oswestry Disability Index (ODI) for Randomisation Arm B | up to 6 weeks
  Oswestry Disability Index is a commonly used scale for back pain subjects with a neuropathic pain component. The test is considered the 'gold standard' of low back functional outcome tools.
Oswestry Disability Index (ODI) for Randomisation Arm C | up to 6 weeks
  Oswestry Disability Index is a commonly used scale for back pain subjects with a neuropathic pain component. The test is considered the 'gold standard' of low back functional outcome tools.
Oswestry Disability Index (ODI) for Randomisation Arm D | up to 6 weeks
  Oswestry Disability Index is a commonly used scale for back pain subjects with a neuropathic pain component. The test is considered the 'gold standard' of low back functional outcome tools.
Oswestry Disability Index (ODI) | At 3 months post randomisation
  Oswestry Disability Index is a commonly used scale for back pain subjects with a neuropathic pain component. The test is considered the 'gold standard' of low back functional outcome tools.
Oswestry Disability Index (ODI) | At 6 months post randomisation
  Oswestry Disability Index is a commonly used scale for back pain subjects with a neuropathic pain component. The test is considered the 'gold standard' of low back functional outcome tools.
Patient Global Impression of Change (PGI-C) for Randomisation arm A | up to 6 weeks
  PGI-C is a standard seven-point scale (1-7) used to assess the SCS outcome. 1= No change, 2= Almost the same, 3=A little better, 4= Somewhat better, 5=Moderately better, 6=Better, 7= A great deal better.
Patient Global Impression of Change (PGI-C) for Randomisation arm B | up to 6 weeks
  PGI-C is a standard seven-point scale (1-7) used to assess the SCS outcome. 1= No change, 2= Almost the same, 3=A little better, 4= Somewhat better, 5=Moderately better, 6=Better, 7= A great deal better.
Patient Global Impression of Change (PGI-C) for Randomisation arm C | up to 6 weeks
  PGI-C is a standard seven-point scale (1-7) used to assess the SCS outcome. 1= No change, 2= Almost the same, 3=A little better, 4= Somewhat better, 5=Moderately better, 6=Better, 7= A great deal better.
Patient Global Impression of Change (PGI-C) for Randomisation arm D | up to 6 weeks
  PGI-C is a standard seven-point scale (1-7) used to assess the SCS outcome. 1= No change, 2= Almost the same, 3=A little better, 4= Somewhat better, 5=Moderately better, 6=Better, 7= A great deal better.
Patient Global Impression of Change (PGI-C) | At 3 Months post randomisation
  PGI-C is a standard seven-point scale (1-7) used to assess the SCS outcome. 1= No change, 2= Almost the same, 3=A little better, 4= Somewhat better, 5=Moderately better, 6=Better, 7= A great deal better.
Patient Global Impression of Change (PGI-C) | At 6 Months post randomisation
  PGI-C is a standard seven-point scale (1-7) used to assess the SCS outcome. 1= No change, 2= Almost the same, 3=A little better, 4= Somewhat better, 5=Moderately better, 6=Better, 7= A great deal better.
EQ-5D 5 Level (EQ-5D-5L) | Baseline
  EQ-5D-5L is comprised of a descriptive system and a visual analogue scale. The descriptive system measures quality of life along five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with five levels for each dimension from which subjects are asked to select one.
EQ-5D 5 Level (EQ-5D-5L) for Randomisation arm A | up to 6 weeks
  EQ-5D-5L is comprised of a descriptive system and a visual analogue scale. The descriptive system measures quality of life along five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with five levels for each dimension from which subjects are asked to select one.
EQ-5D 5 Level (EQ-5D-5L) for Randomisation arm B | Up to 6 weeks
  EQ-5D-5L is comprised of a descriptive system and a visual analogue scale. The descriptive system measures quality of life along five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with five levels for each dimension from which subjects are asked to select one.
EQ-5D 5 Level (EQ-5D-5L) for Randomisation arm C | up to 6 weeks
  EQ-5D-5L is comprised of a descriptive system and a visual analogue scale. The descriptive system measures quality of life along five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with five levels for each dimension from which subjects are asked to select one.
EQ-5D 5 Level (EQ-5D-5L) for Randomisation arm D | up to 6 weeks
  EQ-5D-5L is comprised of a descriptive system and a visual analogue scale. The descriptive system measures quality of life along five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with five levels for each dimension from which subjects are asked to select one.
EQ-5D 5 Level (EQ-5D-5L) | At 3 months post- randomisation
  EQ-5D-5L is comprised of a descriptive system and a visual analogue scale. The descriptive system measures quality of life along five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with five levels for each dimension from which subjects are asked to select one.
EQ-5D 5 Level (EQ-5D-5L) | At 6 months post- randomisation
  EQ-5D-5L is comprised of a descriptive system and a visual analogue scale. The descriptive system measures quality of life along five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with five levels for each dimension from which subjects are asked to select one.
Pain and sleep index 3 (PSQ-3) | Baseline
  PSQ is an eight-item questionnaire developed to assess the impact of pain on quality of sleep. Seven of the eight items are scored using 100 mm VAS, while the remaining item asks individuals to indicate the average number of hours of sleep they get each night. Typically, the first five items on the scale are summed and used as an overall measure of the impact of pain on quality of sleep
Pain and sleep index 3 for Randomisation Arm A | up to 6 weeks
  PSQ is an eight-item questionnaire developed to assess the impact of pain on quality of sleep. Seven of the eight items are scored using 100 mm VAS, while the remaining item asks individuals to indicate the average number of hours of sleep they get each night. Typically, the first five items on the scale are summed and used as an overall measure of the impact of pain on quality of sleep
Pain and sleep index 3 for Randomisation Arm B | up to 6 weeks
  PSQ is an eight-item questionnaire developed to assess the impact of pain on quality of sleep. Seven of the eight items are scored using 100 mm VAS, while the remaining item asks individuals to indicate the average number of hours of sleep they get each night. Typically, the first five items on the scale are summed and used as an overall measure of the impact of pain on quality of sleep
Pain and sleep index 3 for Randomisation Arm C | up to 6 weeks
  PSQ is an eight-item questionnaire developed to assess the impact of pain on quality of sleep. Seven of the eight items are scored using 100 mm VAS, while the remaining item asks individuals to indicate the average number of hours of sleep they get each night. Typically, the first five items on the scale are summed and used as an overall measure of the impact of pain on quality of sleep
Pain and sleep index 3 for Randomisation Arm D | up to 6 weeks
  PSQ is an eight-item questionnaire developed to assess the impact of pain on quality of sleep. Seven of the eight items are scored using 100 mm VAS, while the remaining item asks individuals to indicate the average number of hours of sleep they get each night. Typically, the first five items on the scale are summed and used as an overall measure of the impact of pain on quality of sleep
Pain and sleep index 3 | At 3 months post randomisation
  PSQ is an eight-item questionnaire developed to assess the impact of pain on quality of sleep. Seven of the eight items are scored using 100 mm VAS, while the remaining item asks individuals to indicate the average number of hours of sleep they get each night. Typically, the first five items on the scale are summed and used as an overall measure of the impact of pain on quality of sleep
Pain and sleep index 3 | At 6 months post randomisation
  PSQ is an eight-item questionnaire developed to assess the impact of pain on quality of sleep. Seven of the eight items are scored using 100 mm VAS, while the remaining item asks individuals to indicate the average number of hours of sleep they get each night. Typically, the first five items on the scale are summed and used as an overall measure of the impact of pain on quality of sleep
Pain Drawing | Baseline
  Pain drawing will be used to help patients highlight all the body areas affected by neuropathic pain on a printed dermatome map. It will be collected at the baseline.
Patient Satisfaction with Treatment (PSWT) for Randomisation Arm A | up to 6 weeks
  The Patient Satisfaction with Treatment survey will be used at the end of each Period and at end of study.
Patient Satisfaction with Treatment (PSWT) for Randomisation Arm B | up to 6 weeks
  The Patient Satisfaction with Treatment survey will be used at the end of each Period and at end of study.
Patient Satisfaction with Treatment (PSWT) for Randomisation Arm C | up to 6 weeks
  The Patient Satisfaction with Treatment survey will be used at the end of each Period and at end of study.
Patient Satisfaction with Treatment (PSWT) for Randomisation Arm D | up to 6 weeks
  The Patient Satisfaction with Treatment survey will be used at the end of each Period and at end of study.
Patient Satisfaction with Treatment (PSWT) | At 3 months post randomisation
  The Patient Satisfaction with Treatment survey will be used at the end of each Period and at end of study.
Patient Satisfaction with Treatment (PSWT) | At 6 months post randomisation
  The Patient Satisfaction with Treatment survey will be used at the end of each Period and at end of study.
Electronic pain diary (e-diary) | Up to 7 months
  The patient will be asked to collect information about their pain daily with an e-Diary. A paper version of the diary will be included as a backup if the e-Diary malfunctions or the patient experiences difficulties with the e-Diary recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Mehta, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This study will be registered with the Trust Information Governance Manager at Bart's Health NHS Trust, ensuring the confidentiality of personal data. A signed declaration form (data protection form) of the group to comply with the Data Protection Act and the Department of Health Code of Confidentiality will be applied.

REFERENCES:
- [Background] Kumar K, Hunter G, Demeria D. Spinal cord stimulation in treatment of chronic benign pain: challenges in treatment planning and present status, a 22-year experience. Neurosurgery. 2006 Mar;58(3):481-96; discussion 481-96. doi: 10.1227/01.NEU.0000192162.99567.96. PMID 16528188
- [Background] Owusu S, Huynh A, Gruenthal E, Prusik J, Owusu-Sarpong S, Cherala R, Peng S, Pilitsis JG, McCallum SE. Prospective Evaluation of Patient Usage of Above and Below Threshold Waveforms With Traditional Spinal Cord Stimulation Devices. Neuromodulation. 2017 Aug;20(6):567-574. doi: 10.1111/ner.12633. Epub 2017 Jul 11. PMID 28699301
- [Background] Kapural L, Yu C, Doust MW, Gliner BE, Vallejo R, Sitzman BT, Amirdelfan K, Morgan DM, Brown LL, Yearwood TL, Bundschu R, Burton AW, Yang T, Benyamin R, Burgher AH. Novel 10-kHz High-frequency Therapy (HF10 Therapy) Is Superior to Traditional Low-frequency Spinal Cord Stimulation for the Treatment of Chronic Back and Leg Pain: The SENZA-RCT Randomized Controlled Trial. Anesthesiology. 2015 Oct;123(4):851-60. doi: 10.1097/ALN.0000000000000774. PMID 26218762